CLINICAL TRIAL: NCT07150364
Title: Comparison of Square Stepping Exercise and Wobble Board Exercise on Cognition, Balance and Fall Risk in Elderly Population
Brief Title: Comparison of Square Stepping Exercise and Wobble Board Exercise in Elderly Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/RCR&AHS/24/02101
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Elderly Population
Keywords: Balance; Cognition; Fall risk; Square-stepping exercise; Wobble board

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Square Stepping Exercise (Experimental): In SSE, step patterns are performed on a mat
  Interventions: Other: Square Stepping Exercise
- Wobble Board Exercise (Experimental): Person is standing on a wobble board, that unexpectedly translates or tilts
  Interventions: Other: Wobble Board Exercise

INTERVENTIONS:
Other: Square Stepping Exercise — 5 days per week for 6 weeks. 30 minutes per session with appropriate rest interval in between.
  Arms: Square Stepping Exercise
Other: Wobble Board Exercise — 5 days per week for 6 weeks. 30 minutes per session with appropriate rest interval in between.
  Arms: Wobble Board Exercise

SUMMARY:
Cognitive decline and balance issues are key contributors to falls. Square Stepping Exercise (SSE) and Wobble Board Exercise (WBE) both are the promising forms of balance training. Therefore, the aim of this study is to compare these two exercises to determine their effects on cognition, balance, and fall risk in elderly population.

DETAILED DESCRIPTION:
The study in 2016 described the effects of square stepping exercises versus traditional balance exercises on improving balance and reducing fear of falling in the elderly. The Mini Mental State Examination (MMSE), Berg Balance Scale (BBS), Timed Up and Go (TUG) test, and Fall Efficacy Scale (FES) were used for assessments. Both groups showed significant improvements in BBS and TUG scores (p<0.0001), but the square stepping exercise group demonstrated more significant gains. The study concluded that square stepping exercises were more effective in enhancing balance and reducing fear of falling compared to traditional balance exercises.This study addresses a notable gap in existing literature by comparing the effects of Square Stepping Exercise and Wobble Board Exercise in improving cognition, balance, and fall risk among the elderly. While both exercises have been recognized individually for their benefits, but their comparative effectiveness remains understudied. By focusing on this comparison, this study aim is to fill this gap and offer valuable insights into the most effective intervention for enhancing functional independence and promoting healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals age 60 years and above of both genders according to the guidelines of World Health Organization (WHO).
* Participants whose Mini Mental State Examination (MMSE) score will be >24/30 ensuring sufficient cognitive ability to follow instructions and participate in exercise.
* Participants whose Berg Balance Scale scores of more than 41/56 ensuring that the participants have moderate level of balance ability.
* Vital signs within normal range for elderly population.
* Ability to walk independently with or without an assistive device (e.g., canes).

Exclusion Criteria:

* Participants who have severe musculoskeletal or neurological disorders affecting gait or balance (e.g., Parkinson's disease, and stroke) because of the complex impacts of these conditions on general cognitive and physical functions.
* Participants who undergoes recent fractures or injuries affecting participation in physical activity.
* Participants who have uncontrolled cardiovascular or metabolic conditions (e.g., uncontrolled hypertension, and diabetes mellitus) that could significantly interfere with exercise.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Fall Efficacy Scale- international (FES- I) | 6th week
  The FES-I is designed to assess concern about falling while performing basic and instrumental indoor and outdoor activities. This scale consists of 16 items (10 items from the original FES and six additional social activities items). Each item is scored with a four- point scale (1 = not concerned at all, 4 = very concerned). The summation of scores gives a total score from 16 (absence of FOF) to 64 (extreme concern of falling). This scale was used as a criterion scale in the present study with a cutoff point of 23.
Mini Mental State Examination (MMSE) | 6th week
  The Mini-Mental State Examination (MMSE) is a widely used tool for screening cognitive function and assessing the severity of cognitive impairment. It assesses areas such as orientation, registration, attention and calculation, recall, language, and visual construction. The MMSE consists of 30 questions with a maximum score of 30 points in which score between 24-30 is consider normal, score 18-23 is consider mild cognitive impairment and score between 0-17 is consider severe cognitive impairment.
Berg Balance Scale (BBS) | 6th week
  The BBS evaluates a participant's balance based on 14 items scored and takes 15-20 min to complete. The score for each item ranges from 0 to 4 points, with an overall maximum score of 56 points. Balance is evaluated by asking participants to perform a variety of sitting, transferring and standing positions. In an assessment of which cut- off scores on the BBS best predict the risk of falling. The score of 41-56 indicates low risk of fall, 21-40 indicates medium risk of fall, and 0-20 indicates the high risk of fall.

SECONDARY OUTCOMES:
Time up and Go test (TUG) | 6th week
  The TUG is a performance-based measure of functional mobility initially developed to identify mobility and balance impairments in older adults. The TUG test takes only a few minutes to complete. In this test, participants are asked to stand up from a chair, walk 3 m, turn, walk 3 m back and sit down again. The time taken to perform this task indicates high or low falls risk. The cut- off scores reported in the articles varied from 10.9 seconds to 13 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Tariq, Principal Investigator — Riphah International University
Locations (1):
- Khursheed Old Home, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delbaere K, Valenzuela T, Lord SR, Clemson L, Zijlstra GAR, Close JCT, Lung T, Woodbury A, Chow J, McInerney G, Miles L, Toson B, Briggs N, van Schooten KS. E-health StandingTall balance exercise for fall prevention in older people: results of a two year randomised controlled trial. BMJ. 2021 Apr 6;373:n740. doi: 10.1136/bmj.n740. PMID 33824131
- [Background] Forbes PA, Chen A, Blouin JS. Sensorimotor control of standing balance. Handb Clin Neurol. 2018;159:61-83. doi: 10.1016/B978-0-444-63916-5.00004-5. PMID 30482333
- [Background] Guirguis-Blake JM, Michael YL, Perdue LA, Coppola EL, Beil TL. Interventions to Prevent Falls in Older Adults: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Apr 24;319(16):1705-1716. doi: 10.1001/jama.2017.21962. PMID 29710140
- [Background] Henry M, Baudry S. Age-related changes in leg proprioception: implications for postural control. J Neurophysiol. 2019 Aug 1;122(2):525-538. doi: 10.1152/jn.00067.2019. Epub 2019 Jun 5. PMID 31166819
- [Background] Franzel K, Koschate J, Freiberger E, Shigematsu R, Zieschang T, Tietgen S. Square-stepping exercise in older inpatients in early geriatric rehabilitation. A randomized controlled pilot study. BMC Geriatr. 2024 Apr 10;24(1):326. doi: 10.1186/s12877-024-04932-3. PMID 38600478
- [Background] Thomas E, Battaglia G, Patti A, Brusa J, Leonardi V, Palma A, Bellafiore M. Physical activity programs for balance and fall prevention in elderly: A systematic review. Medicine (Baltimore). 2019 Jul;98(27):e16218. doi: 10.1097/MD.0000000000016218. PMID 31277132
- [Background] Kawabata M, Gan SR, Shen-Hsing AC. Effects of Square Stepping Exercise on cognitive, physical, psychological, and group functioning in sedentary older adults: A center-based hybrid trial. BMC Geriatr. 2024 Apr 25;24(1):374. doi: 10.1186/s12877-024-04904-7. PMID 38664613
- [Background] Taghavi Asl A, Shojaedin SS, Hadadnezhad M. Comparison of effect of wobble board training with and without cognitive intervention on balance, ankle proprioception and jump landing kinetic parameters of men with chronic ankle instability: a randomized control trial. BMC Musculoskelet Disord. 2022 Sep 30;23(1):888. doi: 10.1186/s12891-022-05706-x. PMID 36180870
- [Background] Rudnicka E, Napierala P, Podfigurna A, Meczekalski B, Smolarczyk R, Grymowicz M. The World Health Organization (WHO) approach to healthy ageing. Maturitas. 2020 Sep;139:6-11. doi: 10.1016/j.maturitas.2020.05.018. Epub 2020 May 26. PMID 32747042
- [Background] Meimandi M, Fadavi-Ghaffari M, Taghizadeh G, Azad A, Lajevardi L. Falls Efficacy Scale and Single Item Question: Screening Accuracy for Older Adults Residing in Nursing Homes. Clin Gerontol. 2021 Oct-Dec;44(5):544-551. doi: 10.1080/07317115.2020.1858467. Epub 2020 Dec 15. PMID 33320074
- [Background] Dewan N, MacDermid JC. Fall Efficacy Scale-International (FES-I). J Physiother. 2014 Mar;60(1):60. doi: 10.1016/j.jphys.2013.12.014. Epub 2014 May 3. No abstract available. PMID 24856947
- [Background] Patnode CD, Perdue LA, Rossom RC, Rushkin MC, Redmond N, Thomas RG, Lin JS. Screening for Cognitive Impairment in Older Adults: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2020 Feb 25;323(8):764-785. doi: 10.1001/jama.2019.22258. PMID 32096857
- [Background] Meekes WM, Korevaar JC, Leemrijse CJ, van de Goor IA. Practical and validated tool to assess falls risk in the primary care setting: a systematic review. BMJ Open. 2021 Sep 29;11(9):e045431. doi: 10.1136/bmjopen-2020-045431. PMID 34588228
- [Background] Zahedian-Nasab N, Jaberi A, Shirazi F, Kavousipor S. Effect of virtual reality exercises on balance and fall in elderly people with fall risk: a randomized controlled trial. BMC Geriatr. 2021 Sep 25;21(1):509. doi: 10.1186/s12877-021-02462-w. PMID 34563120